CLINICAL TRIAL: NCT03037996
Title: The Develop a Validated Si-2-AQ and Use it to Evaluate Patients Postoperatively
Brief Title: To Develop a Validated Program and Use it to Evaluate Patients Post-operatively
Acronym: Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Sudta Parakkamodom, Principal Investigator, Siriraj Hospital
Other Study IDs: COA no. Si 790/2016
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Patient Relations, Nurse; Post-operative Patients
Keywords: anesthesia; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients' response — patients' satisfaction to anesthesia services

SUMMARY:
Annually, the Department of Anesthesiology, Siriraj hospital has responsibilities to take care of more than 50,000 patients peri-operatively. According to Maslow's hierarchy of needs; human's pleasure is classified as physiological, safety, belonging, esteem and self-actualization. Since defining and measuring quality of healthcare service is an inevitable challenge for all institutes in medical fields, a questionnaire is developed to assess the quality of all services. The Siriraj Anesthesia Quality Assessment Questionnaire (Si-2-AQ), a simply 40-item tool in seven dimensions, comprises Accessibility and convenience, Communication and Information, Process of care, Technical Quality, Psychological support, Physical support and Royalty.

DETAILED DESCRIPTION:
Anesthesia service is the medical specialty that focuses on peri-operative medicine and the administration of anesthetics. It expresses traditionally as the conditions of no pain perception during surgical procedure. This includes three broad categories: 1) General Anesthesia is a medically induced state of unconsciousness with loss of protective reflexes; 2) Sedation is a state of irritability or agitation reduction to facilitate a medical or diagnostic procedure; and 3) Regional Anesthesia is a technique to abolish either or both motor and sensory sensitivity in a specific part of the body.

Siriraj Hospital, Mahidol University, Bangkok is a tertiary, general hospital with more than 2,200 beds. Annually, the Department of Anesthesiology has responsibilities to take care of more than 50,000 patients peri-operatively. Currently, it plays a part in many surgical departments: Traumatic surgery (TRAU); Orthopedics surgery (ORT); Eye surgery (EYE); Ear, Nose and Throat surgery (ENT); Plastics surgery (PLA); Cardio-thoracic surgery (CVT); Neurosurgery (NEU); General surgery (GEN), Urological surgery (URO); Head and Neck surgery (H&N); Pediatric surgery (PED); Obstetrics surgery (OBG); Gynecological surgery (GYN); Electro-convulsive therapy (PSY); Radiological services (RAD); Endoscopic center (SCOP); Intensive Care Unit (ICU); Acute Pain service (APS); Pain Clinic (PC); and Pre-Anesthesia Assessment Center (SiPAC).

According to Maslow's hierarchy of needs; human's pleasure is classified as physiological, safety, belonging, esteem and self-actualization. Likewise, patients' satisfaction seems to cover all these aspects; since participants crave for an excellent healthcare services. As a result, their contentment become a crucial factor to determine the quality of care particularly in Anesthesia procedure. This includes many processes in peri-Anesthesia management such as patient safety in operating theater, pain controlling and mutually convenient inter-relationship, etc. To solve these procedural running by means of patients' desires, a quality survey seems to be a promising tool that right on the target.

Since defining and measuring quality of healthcare service is an inevitable challenge for all institutes in medical fields, many organizations try to work out intensively. Currently, there are many leading quality assessment tools in healthcare services, namely Hospital Consumer Assessment of Healthcare Providers and System (HCAHPS), Patient Satisfaction Questionnaire (PSQ), Service Quality Questionnaire (SERVQUAL), Quality of Recover after anesthesia 40 (QoR-40), Post-operative Quality of Recovery Questionnaire and Developing and Testing Questionnaire. These tests have been already verified for its validity and reliability.

HCAHPS a 33-item survey in three dimensions, comprises nurse and doctor communication, medical communication, responsiveness of hospital staff, pain management, discharge information, care transition 17 items; cleanliness and quietness of hospital environment 2 items; as well as overall rating of hospital and willingness to recommend hospital 2 items.

PSQ an 18-item questionnaire in seven dimensions, consists of general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor as well as accessibility and convenience.

SERVQUAL a questionnaire related to hospital services in five dimensions, is composed of tangibles, reliability, responsiveness, assurance and empathy.

QoR-40 a 40-item questionnaire concerning good quality recovery after anesthesia and surgery, includes emotional states, physical and physiological support, physical independence and pain management.

Based upon the previously mentioned; investigators, therefore, would like to develop a questionnaire to assess the quality of our services. The Siriraj Anesthesia Quality Assessment Questionnaire (Si-2-AQ), a simply 40-item tool in seven dimensions, comprises Accessibility and convenience (5 items), Communication and Information (10 items), Process of care (8 items), Technical Quality (9 items) Psychological support (4 items) Physical support (2 items) and Royalty (2 items).

ELIGIBILITY:
Inclusion Criteria:

* Volunteered, literate and communicable, well-conscious, in-patients ASA I-III, aged 18-65 years who underwent elective surgery.

Exclusion Criteria:

* Patients with severe diseases such as congestive heart failure, end-stage renal disease, etc. Patients refuse to join the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A developed and validated questionnaire will be studied in 450 patients as target group (4 months). Post-operatively, a nurse anesthetist visits a patient to explain the details of the study and ask for consent. Afterwards, a participant responses to a questionnaire privately (10 minutes). Co-investigators collect data in a computer file. A statistician who not involved in the study analyzes the data.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients' satisfaction | 4 months
  questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Chairal Shayakul, M.D., Study Chair — Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok

IPD SHARING:
Plan to Share IPD: No